CLINICAL TRIAL: NCT05668988
Title: A Phase 3, Open-Label, Randomized, Multi-Center Study of DZD9008 Versus Platinum-Based Doublet Chemotherapy as First-Line Treatment for Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer Harboring Epidermal Growth Factor Receptor Exon 20 Insertion Mutation
Brief Title: A Study of DZD9008 Versus Platinum-Based Doublet Chemotherapy in Local Advanced or Metastatic Non-small Cell Lung Cancer (WU-KONG28)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Dizal Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DZ2022E0005
Record Dates: First submitted 2022-12-20; First posted 2022-12-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-02

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- sunvozertinib (Experimental)
  Interventions: Drug: sunvozertinib
- Platinum-based Chemotherapy (Active Comparator)
  Interventions: Drug: Pemetrexed+carboplatin

INTERVENTIONS:
Drug: sunvozertinib — orally, 300 mg, once daily until a treatment discontinuation criterion is met.
  Arms: sunvozertinib
Drug: Pemetrexed+carboplatin — Participants randomized into chemotherapy arm can receive up to 6 cycles of pemetrexed + carboplatin (pemetrexed 500 mg/m2 + carboplatin area under the plasma concentration-time curve 5 mg/ml per minute (AUC5), IV infusion, every 3 weeks) as the initial treatment. Participants whose disease has not progressed after 4 cycles of first-line platinum-based doublet chemotherapy may receive pemetrexed maintenance monotherapy until a treatment discontinuation criterion is met.
  Arms: Platinum-based Chemotherapy

SUMMARY:
This is a phase 3, open-label, randomized, multi-center study assessing the efficacy and safety of DZD9008 versus platinum-based doublet chemotherapy in participants with locally advanced or metastatic NSCLC with EGFR Exon20ins mutation, who are newly diagnosed or have not received prior systemic therapy in advanced stage.

Primary objective of this study is to assess the efficacy of DZD9008 versus platinum-based doublet chemotherapy using by BICR-assessed PFS per RECIST 1.1 as primary endpoint. Approximately 320 participants are estimated to be randomized into the study. Participants enrolled will be randomized to DZD9008 or platinum-based doublet chemotherapy in a 1:1 manner, stratified by baseline brain metastasis (with/without).

ELIGIBILITY:
Inclusion Criteria:

1. Aged at least 18 years old (or per local regulatory/IRB requirement).
2. Histologically or cytologically confirmed diagnosis of non-squamous NSCLC, locally advanced (Stage IIIB and IIIC according to the 8th edition of the AJCC TNM staging criteria) or metastatic (Stage IV), not suitable for curative therapy.
3. Adequate tumor tissue available, for central laboratory confirmation of EGFR exon 20 insertion mutation
4. At least 1 measurable lesion per RECIST Version 1.1
5. Life expectancy ≥ 12 weeks
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
7. Adequate organ and hematologic function

Exclusion Criteria:

1. Prior treatment with any systemic anti-cancer therapy for locally advanced or metastatic NSCLC.
2. Spinal cord compression or leptomeningeal metastasis.
3. Concurrent EGFR mutations: exon 19 deletion, L858R, T790M, G719X, S768I, or L861Q.
4. History of stroke or intracranial hemorrhage within 6 months before randomization.
5. As judged by the investigator, any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses (i.e., hemophilia and Von Willebrand disease).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Actual)
Dates: Start 2022-12-13 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) as assessed by Blinded Independent Central Review (BICR) per RECIST 1.1 | Up to approximately 34 months after the first participant is randomized

SECONDARY OUTCOMES:
Overall Survival | Up to approximately 34 months after the first participant is randomized

CONTACTS AND LOCATIONS:
Overall Officials: Caicun Zhou, Principal Investigator — Shanghai Pulmonary Hospital, Shanghai, China
Locations (160):
- United States (15):
  - OPN Healthcare, Inc., Glendale, California
  - Kaiser Permanente Medical Center, Vallejo, California
  - University of Colorado Hospital - Anschutz Cancer Pavilion, Aurora, Colorado
  - D&H Cancer Research Center, Margate, Florida
  - Brcr Global, Plantation, Florida
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - NYU Laura & Issac Perlmutter Cancer Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Gabrail Cancer Center Research, Canton, Ohio
  - The Ohio State University, Columbus, Ohio
  - Providence Portland Medical Center, Portland, Oregon
  - USOR - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - MD Anderson cancer center, Houston, Texas
  - USOR - Texas Oncology--Weslaco, Weslaco, Texas
  - University of Virginia Comprehensive Cancer Center, Charlottesville, Virginia
- Argentina (11):
  - Centro de Educación Médica e Investigaciones Clínicas, CEMIC, Buenos Aires
  - Centro Diabaid, Buenos Aires
  - Centro Medico Austral, Buenos Aires
  - Consultorios Medicos Dr. Doreski - Fundacion Respirar, Buenos Aires
  - Fundacion Cenit Para El Estudio De Neurociencias, Buenos Aires
  - Hospital Italiano de Buenos Aires (HIBA), Buenos Aires
  - Instituto Alexander Fleming, Buenos Aires
  - Instituto Argentino de Diagnositco y Tratamiento S.A, Buenos Aires
  - Fundación Estudios Clínicos, Rosario
  - Fundación Ars Médica, San Salvador
  - Centro de Investigación Clínicas. Clinica Viedma S.A, Viedma
- Australia (4):
  - Concord Cancer Centre Medical Oncology Clinical Trials Unit Concord Repatriation General Hospital, Concord
  - Peter MacCallum Cancer Centre, Melbourne
  - Sir Charles Gairdner Hospital, Heart Research Insititute, Nedlands
  - Prince of Wales Hospital, Randwick
- Austria (2):
  - Ordensklinikum Linz GmbH Elisabethinen, Linz
  - Uniklinikum Salzburg, Salzburg
- Belgium (3):
  - Antwerpen University Hospital (UZA), Edegem, Antwerp
  - University Hospital Gent- Drug Research Unit Ghent (D.R.U.G.), Ghent, Flanders
  - Grand Hopital de Charleroi (GHdC) - Hopital Notre Dame, Charleroi, Hainaut
- Brazil (10):
  - Fundacao PIO XII - Hospital do Cancer de Barretos, Barretos
  - Centro de Pesquisas Clinicas em, Cachoeiro de Itapemirim
  - Liga Norte Riograndense Contra o Câncer, Natal
  - Hospital São Lucas da PUCRS, Porto Alegre
  - Santa Casa de Misericordia- Porto Alegre - Hospital Santa Rita, Porto Alegre
  - Instituto D'Or de Pesquisa e Ensino - Recife, Recife
  - Instituto America(COI), Rio de Janeiro
  - Instituto D'Or de Pesquisa e Ensino, Rio de Janeiro
  - Instituto Nacional de Cancer Jose Alencar Gomes da Silva, Rio de Janeiro
  - Instituto do Cancer do Estado de Sao Paulo - ICES, São Paulo
- Canada (3):
  - Regional Cancer Program London Health Sciences Centre, London
  - The Ottawa Hospital Cancer Center, Ottawa
  - Princess Margaret Cancer Center, Toronto
- China (42):
  - Beijing Cancer Hospital, Beijing
  - Beijing Chest Hospital, Capital Medical University, Beijing
  - Cancer Hospital of the Chinese Academy of Medical Sciences, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - Hunan Cancer Hospital, Changsha
  - West China Hospital of Sichuan University, Chengdu
  - Army Medical Center of PLA, Chongqing
  - Chongqing Cancer Hospital, Chongqing
  - Fujian Cancer Hospital, Fuzhou
  - Fujian Medical University Union Hospital, Fuzhou
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou
  - The First Affiliated Hospital Zhejiang University School of Medicine, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Anhui Provincial Hospital, Hefei
  - The First Affiliated Hospital of Anhui Medical University, Hefei
  - The Affiliated Hospital of Inner Mongolia Medical University, Hohhot
  - Jilin Cancer Hospital, Jilin
  - Central Hospital Affiliated to Shandong First Medical University, Jinan
  - Shandong Cancer Hospital & Institution, Jinan
  - Yunnan Cancer Hospital, Kunming
  - The Second Affiliated Hospital of Nanchang University, Nanchang
  - Jiangsu Cancer Hospital, Nanjing
  - Jiangsu Provincial Hospital, Nanjing
  - Guangxi Medical University Cancer Hospital, Nanning
  - Shanghai Chest Hospital, Shanghai
  - Shanghai Pulmonary Hospital, Shanghai
  - ZhongShan Hospital Fudan University, Shanghai
  - The First Hospital of China Medical University, Shenyang
  - Cancer Hospital Chinese Academy of Medical Sciences, ShenZhen center, Shenzhen
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang
  - Shanxi Provincial Cancer Hospital, Taiyuan
  - Taizhou Hospital of Zhejiang Province, Taizhou
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin
  - Tongji Hospital affiliated to Tongji Medical College of Huazhong University of Science & Technology, Wuhan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - The First Affiliated Hospital of Xi 'an Jiaotong University, Xi'an
  - Yantai Yuhuangding Hospital, Yantai
  - Henan Cancer Hospital, Zhengzhou
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou
- Czechia (2):
  - Fakultni Nemocnice Olomouc (FNOL) - Onkologicka Klinika, Olomouc
  - Vitkovicka Nemocnice a.s. - Plicni oddeleni, Ostrava
- France (16):
  - Centre Hospitalier Universitaire d'Angers, Angers
  - Hôpital Louis Pradel, Bron
  - Centre Hospitalier Intercommunal de Creteil (CHIC), Créteil
  - Centre Hospitalier Universitaire de Lille (CHU Lille) - Hopital Albert Calmette - Clinique des Maladies Respiratoires, Hellemmes-Lille
  - Centre Hospitalier Universitaire Grenoble Alpes (CHU Grenoble Alpes) - Hopital Albert Michallon, La Tronche
  - APHM-Hôpital NORD, Marseille
  - Centre de Cancérologie Montpellier, Montpellier
  - APHP Hôpital Tenon, Paris
  - Cochin Hospital, Paris
  - Hopital Saint Joseph, Paris
  - Hôpital Bichat - Claude Bernard, Paris
  - CHU Poitiers, Poitiers
  - Centre Hospitalier Universitaire de Nantes (CHU de Nantes), Saint-Herblain
  - Institut de Cancerologie de L'Ouest, Saint-Herblain
  - Hopital d'Instruction Des Armees Begin, Saint-Mandé
  - Hopital Foch, Suresnes
- Germany (6):
  - Evangelische Lungenklinik Berlin - Klinik fuer Pneumologie, Berlin
  - Asklepios Klinik Gauting GmbH - Klinik fuer Thorakale Onkologie, Gauting
  - Niels-Stensen-Kliniken - Franziskus-Hospital Harderberg, Georgsmarienhütte
  - Universitaetsklinikum Heidelberg (UKHD) - Thoraxklinik-Heidelberg gGmbH, Heidelberg
  - Universitaetsmedizin der Johannes Gutenberg-Universitaet Mainz - III. Medizinische Klinik und Poliklinik, Mainz
  - Pius-Hospital Oldenburg - Klinik fuer Haematologie und Onkologie, Oldenburg
- Italy (14):
  - Centro di Riferimento Oncologico (CRO Aviano), Aviano
  - Azienda Ospedaliero Universitaria di Bologna - Policlinico S. Orsola-Malpighi, Bologna
  - Azienda Ospedaliero - Universitaria "Policlinico-Vittorio Emanuele" Catania, Catania
  - Università degli Studi di Firenze - Azienda Ospedaliero-Universitaria Careggi (AOUC) - SC di Oncologia MedicaI, Florence
  - Azienda USL Toscana Sud Est -Ospedale Misericordia - Grosseto, Grosseto
  - Servizio Sanitario Regionale Emilia-Romagna - Istituto Scientifico Romagnolo per lo Studio e La Cura dei Tumori Srl (IRST), Meldola
  - Azienda Ospedaliero-Universitaria di Modena (AOU Modena) - Policlinico di Modena, Modena
  - Azienda Ospedaliera San Gerardo - Monza, Monza
  - La Maddalena Casa di Cura di Alta Specialita - Palermo, Palermo
  - Azienda Ospedaliero-Universitaria di Parma, Parma
  - Azienda Unità Sanitaria Locale Romagna, Ravenna
  - Azienda Ospedaliera di Reggio Emilia - Arcispedale S. Maria Nuova (ASMN), Reggio Emilia
  - IRCCS Istituti Fisioterapici Ospitalieri- Istituto Nazionale tumori Regina Elena, Roma
  - Azienda Ospedaliera Universitaria Senese - Istituto Toscano Tumori (ITT) - Center for Immuno-Oncology (CIO), Siena
- Universiteit Maastricht (UM) - Maastricht University Medical Centre (Maastricht UMC+), Maastricht, Netherlands
- Poland (4):
  - Uniwersyteckie Centrum Kliniczne, Klinika Onkologii i Radioterapii, Gdansk
  - MED-POLONIA Sp. z o.o., Poznan
  - Wojewódzki Szpital im. św. Ojca Pio, Przemyśl
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie Panstwowy, Warsaw
- Spain (19):
  - Institut Catala d'Oncologia Badalona (ICO Badalona) - Hospital Germans Trias i Pujol, Barcelona, Barcelona
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Instituto Oncológico Dr Rosell Hospital Quiron Dexeus, Barcelona
  - UOMI Cancer Center - Clinica Tres Torres, Barcelona
  - Institut Catala d'Oncologia de Girona -Hospital Universitari Dr Josep Trueta, Girona
  - Hospital Universitario de Jerez, Jerez de la Frontera
  - Clínica Universidad de Navarra - Madrid, Madrid
  - Hospital HM Sanchinarro, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Fundación Jiménez Diaz, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Regional Universitario de Málaga, Málaga
  - Hospital Universitario Virgen de Valme, Seville
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Universitari i Politècnic La Fe, Valencia
- Turkey (Türkiye) (8):
  - Ankara Bilkent City Hospital Universiteler Mahallesi, Ankara
  - Dr. Abdurrahman Yurtaslan Ankara Oncology Training, Ankara
  - Gazi Universitesi Tip Fakultesi (Gazi University Faculty of Medicine) - Gazi Hastanesi (Gazi Hospital), Ankara
  - Liv Hospital Ankara - Medical Oncology Clinic, Ankara
  - Trakya Universitesi Saglik Arastirma ve Uygulama Merkezi Hastane, Edirne
  - Bezmialem University Hospital, Istanbul
  - Prof. Dr. Süleyman Yalçın Şehir Hastanesi - Tibbi Onkoloji Klinigi, Kadıköy
  - Necmettin Erbakan University, Konya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang M, Fan Y, Sun M, Wang Y, Zhao Y, Jin B, Hu Y, Han Z, Song X, Liu A, Tang K, Ding C, Liang L, Wu L, Gao J, Wang J, Cheng Y, Zhou J, He Y, Dong X, Yao Y, Yu Y, Wang H, Sun S, Huang J, Fang J, Li W, Wang L, Ren X, Zhou C, Hu Y, Zhao D, Yang R, Xu F, Huang Y, Pan Y, Cui J, Xu Y, Yang Z, Shi Y. Sunvozertinib for patients in China with platinum-pretreated locally advanced or metastatic non-small-cell lung cancer and EGFR exon 20 insertion mutation (WU-KONG6): single-arm, open-label, multicentre, phase 2 trial. Lancet Respir Med. 2024 Mar;12(3):217-224. doi: 10.1016/S2213-2600(23)00379-X. Epub 2023 Dec 12. PMID 38101437